CLINICAL TRIAL: NCT01711216
Title: A Post-Marketing, Prospective, Multicenter, Observational Program: Treatment Regimen in Menstrual Cycle Regularization and Persistence in Routine Clinical Practice in Russia, Ukraine, Kazakhstan and Uzbekistan
Brief Title: Treatment Regimen in Menstrual Cycle Regularization and Persistence in Routine Clinical Practice in Russia, Ukraine, Kazakhstan and Uzbekistan
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: P13-688
Record Dates: First submitted 2012-08-22; First posted 2012-10-22 (Estimated); Results first posted 2015-10-30 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-11

CONDITIONS: Irregular Menstrual Cycle
Keywords: Dydrogesterone; Irregular Menstrual Cycle; Progestins
MeSH Terms: conditions — Menstruation Disturbances

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- women received dydrogesterone for irregular menstrual cycle: Adult women received dydrogesterone for irregular menstrual cycle as per standard clinical practice of the treating physician

SUMMARY:
Dydrogesterone is approved in more than 100 countries including Russia, Ukraine, Kazakhstan and Uzbekistan and widely used for the treatment of progesterone deficiencies such as for management of dysmenorrhea, endometriosis, secondary amenorrhea, irregular cycles, dysfunctional uterine bleeding, pre-menstrual syndrome, threatened and habitual miscarriage, infertility due to luteal insufficiency, as well as part of hormone replacement therapy. There are limited data regarding dydrogesterone's role in achieving cycle regularization from post-marketing settings. There is need to assess the persistence of dydrogesterone therapy in a post-marketing setting after cessation of treatment and whether the persistence, if any, is related to the duration of dydrogesterone therapy. Hence, in this observational program, the goal is to observe the possible implications of such treatment in terms of treatment length and response pattern.

DETAILED DESCRIPTION:
The program is designed as a prospective, multicentre, observational, non-interventional, non-randomized, non-controlled, single arm, post-marketing program. Being an observational program, the assignment of patients to dydrogesterone therapy will not be decided with an intention to include patients in the program, but will be guided as per standard clinical practice of the treating physician. Hence the prescribing of dydrogesterone will be clearly separate from the decision to include patients in this program. All dydrogesterone prescriptions will be made in accordance with locally approved package insert for dydrogesterone.

ELIGIBILITY:
Inclusion Criteria

* Women aged 18-40 years
* Irregular menstrual cycle due to progesterone deficiency for at least 3 months
* Dydrogesterone prescribed in accordance with locally approved package insert
* Signed written authorization to provide data for the program

Exclusion Criteria

* Known hypersensitivity to the active ingredient or excipients
* Known or suspected progesterone-dependent neoplasms
* Vaginal bleeding of unknown etiology
* Administration of oral contraceptives
* Any other condition that precludes use of dydrogesterone in a particular patient, in accordance with the contraindication, precautions and special warnings listed in the locally approve package insert (for example, patients with rare hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: women with irregular menstrual cycle due to progesterone deficiency
Sampling Method: Non-Probability Sample
Enrollment: 999 (Actual)
Dates: Start 2012-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Pexman-Fieth, MD, Study Director — Abbott
Locations (66):
- Kazakhstan (17):
  - Site reference ID/Investiagor# 82286, Aktobe
  - Site reference ID/Investiagor# 82287, Aktobe
  - Site reference ID/Investigator# 101795, Aktobe
  - Site reference ID/Investigator# 101799, Aktobe
  - Site reference ID/Investigator# 82279, Aktobe
  - Site reference ID/Investigator# 101798, Aktobe
  - Site reference ID/Investiagor# 82281, Almaty
  - Site reference ID/Investigator# 82293, Almaty
  - Site reference ID/Investigator# 101796, Astana
  - Site reference ID/Investigator# 101797, Astana
  - Site reference ID/Investigator# 82277, Astana
  - Site reference ID/Investigator# 82299, Astana
  - Site reference ID/Investigator# 82300, Astana
  - Site reference ID/Investigator# 82301, Astana
  - Site reference ID/Investiagor# 82282, Shymkent
  - Site reference ID/Investigator# 82275, Shymkent
  - Site reference ID/Investigator# 82288, Shymkent
- Russia (19):
  - Site reference ID/Investigaotr# 76702, Irkutsk
  - Site reference ID/Investigator# 77753, Kazan'
  - Site reference ID/Investigaotr# 76704, Kemerovo
  - Site reference ID/Investigator# 76701, Krasnodar
  - Site reference ID/Investigaot# 88537, Moscow
  - Site reference ID/Investigaotr# 76708, Moscow
  - Site reference ID/Investigator# 76700, Moscow
  - Site reference ID/Investigator# 87013, Moscow
  - Site reference ID/Investigaot# 88535, Moscow
  - Site reference ID/Investigaot# 88514, Nizhny Novgorod
  - Site reference ID/Investigator# 83633, Novosibirsk
  - Site reference ID/Investigaot# 88536, Saint Petersburg
  - Site reference ID/Investigaotr# 76709, Saint Petersburg
  - Site reference ID/Investigator# 77754, Saint Petersburg
  - Site reference ID/Investigaotr# 76705, Tomsk
  - Site reference ID/Investigator# 77755, Tyumen
  - Site reference ID/Investigator# 82036, Volgograd
  - Site reference ID/Investigaot# 88513, Voronezh
  - Site reference ID/Investigator# 82035, Yekaterinburg
- Ukraine (13):
  - Site reference ID/Investigaot# 75815, Dnipropetrovsk
  - Site Reference ID/Investigator# 75816, Ivano-Frankivsk
  - Site reference #/Investigator ID 77816, Kharkiv
  - Site reference ID/Investigaot# 75817, Kharkiv
  - Site reference ID/Investigaot# 75813, Kiev
  - Site Reference ID/Investigator# 75814, Kiev
  - Site reference ID/Investigaot# 88056, Lviv
  - Site reference ID/Investigaot# 75819, Mykolaiv
  - Site reference ID/Investigaot# 77817, Odesa
  - Site reference ID/Investigaot# 80193, Odesa
  - Site reference ID/Investigator # 77813, Ternopil
  - Site reference ID/Investigaot# 75818, Vinnytsia
  - Site Reference ID/Investigator# 75822, Zaporizhzhia
- Uzbekistan (17):
  - Site reference ID/Investigaot# 91973, Andijan
  - Site reference ID/Investigaot# 91974, Andijan
  - Site reference ID/Investigaot# 91987, Bukhara
  - Site reference ID/Investigaot# 91975, Fergana
  - Site reference ID/Investigaot# 91986, Samarkand
  - Site reference ID/Investigaot# 100616, Tashkent
  - Site reference ID/Investigaot# 91984, Tashkent
  - Site reference ID/Investigaot# 91977, Tashkent
  - Site reference ID/Investigaot# 91981, Tashkent
  - Site reference ID/Investigaot# 91982, Tashkent
  - Site reference ID/Investigaot# 92473, Tashkent
  - Site reference ID/Investigaot# 91988, Tashkent
  - Site reference ID/Investigaot# 92474, Tashkent
  - Site reference ID/Investigaot# 91976, Tashkent
  - Site reference ID/Investigaot# 91983, Tashkent
  - Site reference ID/Investigaot# 91980, Urgench
  - Site reference ID/Investigaot# 91985, Urgench

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1000 patients were screened. 1 Patient failed screening and 999 were enrolled into the program.
Period: Overall Study
Arm/Group | Women Received Dydrogesterone for Irregular Menstrual Cycle
Started | 999
Completed | 782
Not Completed | 217
Not completed — Adverse Event | 4
Not completed — Pregnancy | 56
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 46
Not completed — variety of other minor reasons | 83
Not completed — no reason specified | 22

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All eligible patients who received at least 1 dose of program drug and at most 6 treatment cycles
Arm/Group | Women Received Dydrogesterone for Irregular Menstrual Cycle
Number analyzed (Participants) | 955
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.3 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 955
  Male | 0
Region of Enrollment [Number; unit: participants]
  Russian Federation | 382
  Ukraine | 284
  Uzbekistan | 160
  Kazakhstan | 129

OUTCOME MEASURES:

1. Secondary Outcome: Proportion of Patients Reporting at Least One Regular Cycle Over the Treatment Period
Description: Regular cycle is defined as cycle duration between 21 to 35 days, inclusive. Treatment period in this observational program can be from 1 cycle to 6 consecutive cycles. This program does not include patients who required dydrogesterone therapy, according to physician's decision, more than 6 consecutive cycles
Time Frame: Up to 6 months
Population: as for baseline characteristics
Measure: Number; unit: percentage of subjects
Arm/Group | Women Received Dydrogesterone for Irregular Menstrual Cycle
Number analyzed (Participants) | 955
percentage of subjects | 99.1

2. Secondary Outcome: Change of Cycle Duration From Baseline to End of Treatment in Days in Group of Patients With Polymenorrhea
Description: Polymenorrhea was defined as cycle duration < 21 days and the change in duration of the menstrual cycle during treatment was evaluated
Time Frame: From 1 month to 6 months
Population: Full Analysis Set (FAS): All eligible patients who received at least 1 dose of program drug and at most 6 treatment cycles. Patients with polymenorrhoea in FAS
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Women Received Dydrogesterone for Irregular Menstrual Cycle
Number analyzed (Participants) | 109
days | 4.9 (5.9)

3. Secondary Outcome: Change of Cycle Duration From Baseline to End of Treatment in Days in Group of Patients With Oligomenorrhea
Description: Oligomenorrhea is defined as cycle duration > 35 days and the change in duration of the menstrual cycle during treatment was evaluated
Time Frame: From 1 month to 6 months
Population: Full Analysis Set (FAS): All eligible patients who received at least 1 dose of program drug and at most 6 treatment cycles. Patients with oligomenorrhoea in FAS
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Women Received Dydrogesterone for Irregular Menstrual Cycle
Number analyzed (Participants) | 711
days | -15.7 (19.8)

4. Secondary Outcome: Change of Duration of Menstrual Bleeding in Group of Patients With Polymenorrhea
Description: Polymenorrhea is defined as cycle duration < 21 days and the duration of menstrual bleeding was evaluated from baseline to end of treatment in days
Time Frame: From 1 month to 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Women Received Dydrogesterone for Irregular Menstrual Cycle
Number analyzed (Participants) | 110
days | -1.7 (2.5)

5. Secondary Outcome: Change of Duration of Menstrual Bleeding in Group of Patients With Oligomenorrhea
Description: Oligomenorrhea is defined as cycle duration > 35 days and the duration of menstrual bleeding was evaluated from baseline to end of treatment in days
Time Frame: From 1 month to 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Women Received Dydrogesterone for Irregular Menstrual Cycle
Number analyzed (Participants) | 721
days | -1.4 (2.0)

6. Secondary Outcome: Change of Pain Intensity During Menstruation From Baseline to End of Treatment
Description: Pain intensity will be measured using 11-point Likert scale where 0 means no pain and 10 means worst pain
Time Frame: From 1 month to 6 months
Population: Full Analysis Set (FAS): All eligible patients who received at least 1 dose of program drug and at most 6 treatment cycles. Data from 39 patients missing
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Women Received Dydrogesterone for Irregular Menstrual Cycle
Number analyzed (Participants) | 916
units on a scale | -2.8 (2.8)

7. Secondary Outcome: Change of Intensity of Anxiety From Baseline to the End of Treatment
Description: Intensity of anxiety will be measured using 11-point scale where 0 means no anxiety and 10 means maximum anxiety
Time Frame: From 1 month to 6 months
Population: Full Analysis Set (FAS): All eligible patients who received at least 1 dose of program drug and at most 6 treatment cycles. Data for 51 patients missing.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Women Received Dydrogesterone for Irregular Menstrual Cycle
Number analyzed (Participants) | 904
units on a scale | -2.7 (2.8)

8. Secondary Outcome: Patient Satisfaction With the Treatment
Description: Patient satisfaction will be determined based on a 5-point Clinical Global Impression of Severity scale, where 1 = very dissatisfied, 2 = dissatisfied, 3 = somewhat satisfied, 4 = satisfied, 5 = very satisfied.
Time Frame: Up to 6 months
Population: Full Analysis Set (FAS): 955 patients. All eligible patients who received at least 1 dose of program drug and at most 6 treatment cycles. Data for 36 patients were missing. Therefore, 919 patients were analyzed.
Measure: Number; unit: participants
Arm/Group | Women Received Dydrogesterone for Irregular Menstrual Cycle
Number analyzed (Participants) | 919
participants
  Very satisfied | 288
  satisfied | 568
  somewhat satisfied | 55
  dissatisfied | 7
  very dissatisfied | 1

9. Secondary Outcome: Overall Clinical Response on Treatment Assessed by Physician
Description: Overall clinical response assessed by physician will be determined based on a four-point-scale, where 4 = excellent, 3 = good, 2 = fair, and 1 = poor response.
Time Frame: Up to 6 months
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Women Received Dydrogesterone for Irregular Menstrual Cycle
Number analyzed (Participants) | 919
participants
  excellent | 320
  good | 499
  fair | 90
  poor | 10

10. Secondary Outcome: Proportion of Patients With 3 Consecutive Regular Cycles Out of Total Number of Patients Who Had Achieved Cycle Regularization at the End of Treatment Period
Description: Measured only for patients who had achieved cycle regularization at the end of treatment period. Regular cycle is defined as cycle duration 21-35 days, inclusive
Time Frame: Up to 9 months
Population: Follow-up Analysis Set (subset of FAS): Patients in the FAS for whom the last reported menstrual cycle during the treatment period was regular. Data for 55 patients was missing.
Measure: Number; unit: percentage of subjects
Arm/Group | Women Received Dydrogesterone for Irregular Menstrual Cycle
Number analyzed (Participants) | 860
percentage of subjects
  yes | 91.7
  no | 8.3

11. Secondary Outcome: Proportion of Patients With 6 Consecutive Regular Cycles Out of Total Number of Patients Who Had Achieved Cycle Regularization at the End of Treatment Period
Description: as for outcome 10
Time Frame: Up to 12 months
Population: as for outcome 10
Measure: Number; unit: percentage of subjects
Arm/Group | Women Received Dydrogesterone for Irregular Menstrual Cycle
Number analyzed (Participants) | 860
percentage of subjects
  yes | 78.5
  no | 21.5

12. Secondary Outcome: Change of Duration of Menstrual Bleeding in Days in Group of Patients With Polymenorrhea
Description: Measured only for patients who had achieved cycle regularization at the end of treatment period. Polymenorrhea is defined as cycle duration < 21 days
Time Frame: From 1 month to 12 months
Population: Follow-up Analysis Set (subset of FAS): Patients in the FAS for whom the last reported menstrual cycle during the treatment period was regular. Patients with polymenorrhea in subset of FAS.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Women Received Dydrogesterone for Irregular Menstrual Cycle
Number analyzed (Participants) | 103
days | -0.0 (1.2)

13. Secondary Outcome: Change of Duration of Menstrual Bleeding in Days in Group of Patients With Oligomenorrhea
Description: Measured only for patients who had achieved cycle regularization at the end of treatment period. Oligomenorrhea is defined as cycle duration > 35 days
Time Frame: From 1 month to 12 months
Population: Follow-up Analysis Set (subset of FAS): Patients in the FAS for whom the last reported menstrual cycle during the treatment period was regular. Patients with oligomenorrhea in subset of FAS.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Women Received Dydrogesterone for Irregular Menstrual Cycle
Number analyzed (Participants) | 651
days | 0.1 (1.1)

14. Secondary Outcome: Change of Pain Intensity During Menstruation
Description: Measured only for patients who had achieved cycle regularization at the end of treatment period. Pain intensity will be measured using 11-point Likert scale where 0 means no pain and 10 means worst pain
Time Frame: From 1 month to 12 months
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Women Received Dydrogesterone for Irregular Menstrual Cycle
Number analyzed (Participants) | 860
units on a scale | -0.3 (1.8)

15. Secondary Outcome: Change of Intensity of Anxiety
Description: Will be measured only for patients who had achieved cycle regularization at the end of treatment period. Intensity of anxiety will be measured using 11-point scale where 0 means no anxiety and 10 means maximum anxiety
Time Frame: From 1 month to 12 months
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Women Received Dydrogesterone for Irregular Menstrual Cycle
Number analyzed (Participants) | 860
units on a scale | -0.1 (1.7)

16. Primary Outcome: Number of Patients Received Dydrogesterone Therapy Cycles (by Cycle Number)
Time Frame: up to 6 months
Population: Follow-up analysis set 915 patients. Follow-up Analysis Set (subset of FAS): Patients in the FAS for whom the last reported menstrual cycle during the treatment period was regular. Data for 55 patients was missing. Therefore, 860 patients were analyzed.
Measure: Number; unit: participants
Arm/Group | Women Received Dydrogesterone for Irregular Menstrual Cycle
Number analyzed (Participants) | 860
participants
  1 therapy cycle | 1
  2 therapy cycles | 4
  3 therapy cycles | 269
  4 therapy cycles | 66
  5 therapy cycles | 53
  6 therapy cycles | 467

17. Primary Outcome: Number of Patients With Regular Menstrual Cycles During Follow-up (by Number of Cycles)
Time Frame: up to 6 months
Population: as for outcome 16
Measure: Number; unit: participants
Arm/Group | Women Received Dydrogesterone for Irregular Menstrual Cycle
Number analyzed (Participants) | 860
participants
  0 regular cycles | 6
  1 regular cycle | 32
  2 regular cycles | 31
  3 regular cycles | 29
  4 regular cycles | 26
  5 regular cycles | 56
  6 regular cycles | 545
  7 regular cycles | 84
  8 regular cycles | 40
  9 regular cycles | 11
Statistical Analysis 1: Comparison: Women Received Dydrogesterone for Irregular Menstrual Cycle; Test of association between the number of regular menstrual cycles during the follow-up period and the number of dydrogesterone therapy cycles received during the treatment period (Follow-up Analysis Set) Follow-up Analysis Set (N=915); Test type: Superiority or Other; p = 0.3181, Mantel Haenszel — Test statistic (d.f.) 1.0157 (1) A Mantel-Haenszel chi-square test was used, exact p-value was computed using Monte Carlo estimation

18. Secondary Outcome: Time to Relapse
Description: The intention was to measure time to relapse, but since a regular cycle was maintained longer than the period of follow up observation, no resulting variable counted in time was received. Instead, what was measured was the percentage of participants who maintained a regular cycle. Measured only for patients who had achieved cycle regularization at the end of treatment period.
Time Frame: Up to 6 months or longer after ended treatment
Population: Follow-up Analysis Set (subset of FAS): Patients in the FAS for whom the last reported menstrual cycle during the treatment period was regular. Data for 55 patients was missing.
  Among the patients who achieved cycle regularization (Follow-up Analysis Set), a majority (>85%) maintained regular cycles for the whole follow-up period
Measure: Number; unit: percentage of subjects
Arm/Group | Women Received Dydrogesterone for Irregular Menstrual Cycle
Number analyzed (Participants) | 860
percentage of subjects | 85

ADVERSE EVENTS:
Time Frame: Safety was monitored by recording of serious adverse events (SAEs) and pregnancies and spontaneously reported adverse events (AEs) from signed informed consent up to 30 days after the final dose of dydrogesterone.
Arm/Group | Women Received Dydrogesterone for Irregular Menstrual Cycle
Serious Adverse Events (participants affected / at risk) | 2/986
Other Adverse Events (participants affected / at risk) | 14/986
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Women Received Dydrogesterone for Irregular Menstrual Cycle (N=986)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 (1) — no reasonable possibility of a relationship to the program drug.
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) — no reasonable possibility of a relationship to the program drug.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Women Received Dydrogesterone for Irregular Menstrual Cycle (N=986)
Metrorrhagia (Reproductive system and breast disorders) | 4 (5) — The most commonly reported preferred term
Bronchitis (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Breast pain (Reproductive system and breast disorders) | 2 (2)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (3)
Ovarian cyst (Reproductive system and breast disorders) | 2 (2)
Uternine polyp (Reproductive system and breast disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Follow up period was limited to 6 months of observation. Pregnancy incidence was not the aim of research, however, spontaneous pregnancies were observed in 56 (5.6%) patients following standard dosages of dydrogesterone for irregular cycle treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator shall not publish/present the results without Abbott's prior written consent. In the event that applicable law permits Investigator to publish or present results without Abbott's prior written consent, Investigator shall provide Abbott with a complete copy of such publication or presentation at least 60 days prior to submission for publication or presentation and Investigator shall reasonably consider all comments which Abbott may provide regarding such publication or presentation